CLINICAL TRIAL: NCT03237247
Title: Role of Complete Blood Picture in Predicting the Etiology of Extrahepatic Cholestasis
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Wael M Sayed, principle investigator, Assiut University
Other Study IDs: 17100256
Record Dates: First submitted 2017-07-22; First posted 2017-08-02 (Actual); Last update posted 2017-08-08 (Actual); Status verified 2017-08

CONDITIONS: Extrahepatic Cholestasis
Keywords: extrahepatic cholestasis, CBC
MeSH Terms: conditions — Cholestasis, Extrahepatic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (5):
- Benign: cases with benign biliary stricture
- Calcular OJ: cases with calcular extrahepatic cholestasis
- Malignant Distal: cases with malignant distal extrahepatic cholestasis
- Malignant Proximal: cases with malignant proximal extrahepatic cholestasis
- Intrahepatic: cases with intrahepatic cholestasis

SUMMARY:
Cases with extrahepatic cholestasis are common and faced during day to day clinical practice, however reaching the final etiology is sometimes challenging and needs investigations which are usually expensive, may carry hazards to the patients, or inaccessible so we are in need for a method which is easily available, affordable and safe for aiding in the differential diagnosis of extrahepatic cholestasis. our study aiming to evaluate the role of complete blood count in predicting the etiology of extrahepatic cholestasis.

DETAILED DESCRIPTION:
Extrahepatic cholestasis has various etiologies including benign causes (benign stricture, chronic pancreatitis, choledochal cyst, mirizzi syndrome, etc...), choledocholithiasis, malignant causes (cancer pancreas, gallbladder cancer, cholangiocarcinoma, etc....), parasitic infestations (fasciola hepatica, ascaris lumbricoides, etc......) and other causes. it is essential to detect the exact cause of extrahepatic cholestasis in order to determine treatment options. diagnosing such conditions depends on clinical examination, laboratory investigations, imaging studies, endoscopic procedures, biopsy and even surgical intervention. some of these investigations are expensive, not available, or carry risk to the patients. moreover non of them is accurate 100%. Complete blood count is already available, easy to obtain, not invasive investigation. In these study we are trying to evaluate the role of complete blood count parameters namely RDW, MPV, PDW, PCT, NLR, PLR in the differential diagnosis of extrahepatic cholestasis.

ELIGIBILITY:
Inclusion Criteria:

* patients with extrahepatic cholestasis

Exclusion Criteria:

* age under 14 years
* previous bilio-pancreatic interventions
* hemoglobinopathy
* splenomegaly
* myeloproliferative disorders
* diabetes mellitus
* recent blood transfusion in less than one month

Min Age: 14 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: patients with extrahepatic cholestasis
Sampling Method: Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2017-02-28 (Actual); Study Completion 2017-02-28 (Actual)

PRIMARY OUTCOMES:
differential diagnosis of extrahepatic cholestasis | 10 days
  complete blood count parameters